CLINICAL TRIAL: NCT01590043
Title: Identifying Saliva Markers in Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: LSA002-HMO-CTIL
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-07

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole saliva

GROUPS / COHORTS (3):
- Control: Healthy 3-18 years old participants
  Interventions: Other: Salivary samples
- Inflammatory bowel disease: 3-18 years old patients identified with inflammatory bowel disease
  Interventions: Other: Salivary samples
- Abdominal pain: 3-18 years old patients suffering from abdominal pain not related to Inflammatory bowel disease
  Interventions: Other: Salivary samples

INTERVENTIONS:
Other: Salivary samples — Each participant will give a sample of saliva through spitting for 5 minutes in a sterile tube.
  Other Names: Salivary Analysis

SUMMARY:
Under normal conditions intestinal mucosa presents a baseline "physiological inflammation" caused by a controlled immune response that eliminates offending dietary and microbial antigens. This inflammation disappears once the cause is eradicated. In case of inappropriate immunological response, the inflammation becomes chronic and harmful, resulting in anatomical and functional abnormalities, namely inflammatory bowel disease (IBD).

Although it is critical for the IBD patients to undergo early diagnosis and management before the development of severe complications, but as IBD has vague and non-pathognomonic clinical features, the clinician is usually mislead into late suspicion and detection of IBD.

Diagnosis traditionally depended on a combination of pathologic evaluation together with the histological, clinical, radiological, endoscopic, surgical, laboratory (serological) features. Recently, serological markers were identified and became of special interest as they do not only detect the occurrence of IBD but also the potential of its development and may be used as prognostic tools. More recently, stool markers were detected and used for diagnosis.

Up to now, the market is still lacking a definitive, simple and non-invasive diagnostic tool. Saliva can present an alternative form of body fluids that simplify diagnostic procedures.

Our hypothesis is that IBD patients have special salivary biomarkers that may be identified through salivary analysis, where later on a simple non-invasive test can be applied in the form of an easy-to-use kit, being available at the clinician's clinic for the establishment of an immediate and early diagnosis of the destructive inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Identified with inflammatory bowel disease

Exclusion Criteria:

* medically compromised children
* congenital syndromes
* children on medication chronically or on the day of the examination
* children treated with radiotherapy or chemotherapy.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients identified with infalmmatory bowel disease
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Moti Moskovitz, DMD, PhD, Principal Investigator — Hadassah Medical Organization; Eyal Shteyer, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Palmon R, Brown SJ, Abreu MT. What is the role and significance of serum and stool biomarkers in the diagnosis of IBD? Inflamm Bowel Dis. 2008 Oct;14 Suppl 2:S187-9. doi: 10.1002/ibd.20714. PMID 18816678